CLINICAL TRIAL: NCT01304264
Title: Comparison of Intraocular Pressure, Blood Pressure, Ocular Perfusion and Blood Flow Fluctuations During the Addition of Dorzolamid vs Timolol in Glaucoma Subjects Treated With Prostaglandin Analogue Monotherapy
Brief Title: Intraocular Pressure, Blood Pressure, Ocular Perfusion and Blood Flow Fluctuations in Glaucoma Patients
Status: Completed | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Indiana University School of Medicine (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ingrida Januleviciene, MD, Lithuanian University of Health Sciences
Other Study IDs: 37552
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Open Angle Glaucoma
Keywords: glaucoma, ocular, blood flow, fluctuations
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: No biospecimens will be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- combination topical glaucoma treatment: timolol or dorzolamide add on latanoprost monotherapy
  Interventions: Device: Color Doppler Imaging

INTERVENTIONS:
Device: Color Doppler Imaging — Color Doppler imaging (CDI) system for measurements of blood flow in the ophthalmic (OA), central retinal (CRA), and nasal (NPCA) and temporal (TPCA) posterior ciliary arteries. In each vessel, peak systolic velocity (PSV) and end diastolic velocity (EDV) were determined, and Pourcelot's resistive index will be calculated (RI = (PSV-EDV)/PSV).
  Other Names: timololum maleate; dorzolamidum; latanoprostum

SUMMARY:
To evaluate whether add-on to prostaglandin therapy with twice a day (bid) dorzolamide is statistically superior to twice a day (bid) timolol with regard to increasing ocular blood flow

DETAILED DESCRIPTION:
Hypotensive treatments for glaucomatous optic neuropathy (GON), depending on their chemical composition can influence the ocular circulation independent of intraocular pressure (IOP) reduction. It is therefore important not only to identify ocular blood flow deficits in GON, but also document the influence of GON treatments on the ocular circulation

ELIGIBILITY:
Inclusion Criteria:

* Open angle glaucoma subjects receiving prostaglandin monotherapy in both eyes

Exclusion Criteria:

* younger than 18 years old
* women of child bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Regular visitors of Eye Clinic of Lithuania University of Health Science hospital
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Ocular Color Doppler Imaging | 8 AM; 8 PM
  Color Doppler Imaging
  * Nasal post ciliary artery (NPCA)
  * Temporal posterior ciliary artery (TPCA)
  * Ophthalmic artery (OA)
  * Central retinal artery (CRA)

SECONDARY OUTCOMES:
IOP, BP, OPP (mean, fluctuations, amplitude) | 8 AM-12AM-4PM-8PM
  IOP, BP, OPP (mean, fluctuations, amplitude) Goldmann applanation tonometry Brachial artery pressure and radial pulse

CONTACTS AND LOCATIONS:
Overall Officials: Ingrida Januleviciene, MD, Principal Investigator — Lithuania University of Health Science
Locations (1):
- Eye Clinic Lithuania Health Science Hospital Kaunas Clinics, Kaunas, Lithuania